CLINICAL TRIAL: NCT06773884
Title: Population-based Registry Study on Primary Hip Fracture Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Örebro County (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EPM 2024-03060-01
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Hip Fracture
Keywords: Hip Fracture; Primary Hip Fracture Surgery; Perioperative Risk Factors; Reoperation Rates; Mortality; Geriatric Fractures; Epidemiology; Swedish Perioperative Registry (SPOR); Population-Based Study
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: "Observational Analysis of Primary Hip Fracture Surgery Outcomes" — This study examines outcomes following standard primary hip fracture surgery by analyzing retrospective data from national health registries. The focus is on identifying perioperative and patient-related risk factors that influence outcomes such as reoperation rates, mortality, and secondary fractures within one year of surgery. No experimental or new intervention is introduced in this study.

SUMMARY:
This study aims to describe primary hip fracture surgeries and to identify patient-related and perioperative risk factors affecting outcomes. It will utilize data from the Swedish Perioperative Registry (SPOR) and the Swedish National Patient Register to track epidemiological changes, treatment outcomes, and perioperative factors.

DETAILED DESCRIPTION:
Hip fractures, a significant health concern among the elderly, necessitate hospitalization and surgical intervention, with high mortality and morbidity rates within the first year post-surgery. The study will retrospectively analyze records of approximately 90,000 patients over 18 who underwent hip fracture surgery between 2018 and 2022. Key factors such as age, sex, preoperative health status, and perioperative care methods will be evaluated to determine their impact on complications, reoperation rates, and survival.

This research could inform future clinical practices and policies, aiming to optimize the treatment and management of elderly patients with hip fractures.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 18+ with hip fractures, identified through ICD code S72*, who underwent surgery during the study period.

Exclusion Criteria:

* Patients without a Swedish personal identification number, as this is necessary to link data across registers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who underwent hip fracture surgery and were recorded in SPOR from January 1, 2018, to December 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 90000 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of reoperation and secondary fractures. | One year post-surgery
  Rate of reoperation and secondary fractures within one year post-surgery.

SECONDARY OUTCOMES:
Mortality rate, hospitalization duration, and time to surgery | One year post-surgery
  Mortality rate, hospitalization duration, and time to surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Universitetsjukhuset, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No